CLINICAL TRIAL: NCT06422273
Title: Prophylactic Use of Tranexamic Acid Versus Saline to Prevent Bleeding During Transbronchial Biopsy in Lung Transplant Recipients- A Randomized Double-Blind Trial (Protest Trial)
Brief Title: Protest Trial: TXA vs Saline
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Corewell Health West (Other)
Responsible Party: Principal Investigator, Sheila Krishnan, Principle Investigator, Corewell Health West
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2024-0552
Record Dates: First submitted 2024-05-10; First posted 2024-05-20 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Lung Transplant; Complications Surgical
MeSH Terms: interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The study design will be a single-center, randomized, double-blinded, placebo-controlled study. The control group will receive topical saline (placebo) and the experimental treatment group will receive topical Tranexamic acid (TXA active drug).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The investigational pharmacist will be responsible for randomizing on the day of bronchoscopy to placebo or Tranexamic acid in a 1:1 fashion using REDCap software. The pharmacist will be the only individual aware of the randomization assignment. All other study personnel will be blinded to the randomization assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TXA (Experimental): Tranexamic acid used prophylactically prior to performing transbronchial biopsies in lung transplant recipients.
  Interventions: Drug: Tranexamic Acid
- Saline (Placebo Comparator): Topical Saline (placebo) administered as endobronchial topical application.
  Interventions: Other: Saline (placebo)

INTERVENTIONS:
Drug: Tranexamic Acid — Endobronchial (topical) tranexamic acid used prophylactically prior to performing transbronchial biopsies in lung transplant recipients
  Arms: TXA
Other: Saline (placebo) — Topical Saline (placebo) administered as endobronchial topical application prior to performing transbronchial biopsies in lung transplant recipients.
  Arms: Saline

SUMMARY:
To determine if endobronchial (topical) tranexamic acid used prophylactically prior to performing transbronchial biopsies in lung transplant recipients reduces bleeding risk.

DETAILED DESCRIPTION:
Tranexamic acid (TXA) is an antifibrinolytic agent. It forms a reversible complex that displaces plasminogen from fibrin resulting in inhibition of fibrinolysis. It also inhibits proteolytic activity of plasmin. TXA is frequently used in clinical practice and can be administered via multiple delivery methods, including intravenous, nebulized, and topical. It has been shown to reduce blood loss in a variety of clinical settings without significant adverse effects. It has also been evaluated for prophylactic use with mixed results in reducing bleeding. In our current general pulmonary practice, topical TXA is used variably by pulmonologists during bronchoscopy for post-biopsy bleeding or pulmonary hemorrhage.

The purpose of this research study is to determine if prophylactic topical TXA can reduce bleeding risk in lung transplant patients who undergo transbronchial biopsies. A finding of reduced bleeding would be significant as it could improve clinical outcomes, allow for improved diagnostic yield of biopsy samples, and improve patient experience. It therefore has the potential to change clinical practice and standardize bronchoscopy procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Single or double lung transplant recipients
2. Patients >18 years old
3. Willingness and ability to sign an informed consent for study participation

Exclusion Criteria:

1. Platelet count (<50k/uL)
2. INR (>1.6)
3. Active bleeding
4. Decompensated liver disease
5. History of uremic bleeding or BUN >50
6. Severe pulmonary hypertension (mean PA pressure >40 mmHg on RHC or estimated PA systolic pressure >62 mmHg on TTE within one year of procedure)
7. Known bleeding disorder
8. Allergy to TXA
9. Prior history of severe TBBx-related airway bleeding requiring admission or advanced maneuvers for hemostasis (examples including intubation, bronchial artery embolization, surgical intervention)
10. Contraindications to topical TXA
11. Pregnancy
12. Vulnerable populations
13. Adults of limited English proficiency/non-English speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Bleeding Risk | up to 1 hour
  Bleeding severity will be documented in the following categories: none, mild, moderate, severe and massive

SECONDARY OUTCOMES:
Procedure time Reduction | up to 1 hour
  Procedure times will be recorded for both the tranexamic acid and the control saline group.
Greater yield in tissue samples | up to 1 hour
  This will be measured by the number of pieces of tissue from the pathology report

CONTACTS AND LOCATIONS:
Locations (1):
- Corewell Health Hospitals, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT06422273/Prot_SAP_000.pdf